CLINICAL TRIAL: NCT00668785
Title: Intravitreal Ranibizumab to Treat Macular Edema After Panretinal Photocoagulation (Phase II)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to low enrollment
Sponsor: Jumper, J. Michael, M.D. (Individual)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, J. Michael Jumper, MD, Principal Investigator, Jumper, J. Michael, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3848s
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Proliferative Diabetic Retinopathy; Macular Edema
Keywords: Ranibizumab; Proliferative Diabetic Retinopathy; Macular Edema following Panretinal Photocoagulation; Safety and Efficacy; Intravitreal Injection
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Experimental): Ranibizumab is being used off-label to test the safety and efficacy of its use in Diabetic Macular Edema post panretinal photocoagulation. Ranibizumab 0.5mg at baseline and then again at 30 days and/or 60 days after PRP as deemed appropriate by the Investigator.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — Ranibizumab 0.5mg at baseline and then again at 30 days and/or 60 days after PRP as deemed appropriate by the Investigator.
  Other Names: Lucentis

SUMMARY:
This is a randomized, open-label Phase II study evaluating the safety and efficacy of intravitreally administered ranibizumab 0.5mg in subjects with Proliferative Diabetic Retinopathy experiencing post- Panretinal Photocoagulation (PRP) macular edema.

DETAILED DESCRIPTION:
Levels of VEGF are elevated in eyes wth Diabetic Macular Edema and the expression of VEGF was found to be elevated temporarily following the photocoagulation of human Retinal Pigment Epithelial (RPE) cells. Ranibizumab (Lucentis TM, Genentech) is an anti-VEGF antibody shown to have properties to prevent macular edema. We hypothesize that VEGF inhibition can effectively treat PRP-induced macular edema, thereby minimizing post-PRP vision loss.

Subjects who meet eligibility criteria will receive 0.5mg ranibizumab administered 7-14 days post-PRP. Additional intravitreal injections of 0.5 mg of ranibizumab at Day 30 and/or Day 60 may be also be administered. All subjects will be followed for 90 days for safety and efficacy assessments. There is no placebo or sham arm of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Pre-PRP protocol refraction, fluorescein angiography, and optical coherence tomography AND 7-14 day post-PRP OCT
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 21 years or older
* Previously untreated PDR patients with high risk characteristics who develop edema within 7-14 days post PRP therapy. This edema, determined by a masked investigator, will be characterized as either increased foveal thickness (>10% increase from pre-PRP foveal thickness), and/or increased macular volume on OCT (>10% increase from pre-PRP macular volume).

Exclusion Criteria:

* Pregnancy (positive pregnancy test) prior to enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in another simultaneous medical investigation or trial
* Pre-PRP clinically significant diabetic macular edema (CSME) that would make the patient eligible for macular laser prior to PRP
* Neovascularization of the iris or neovascular glaucoma
* Increased central foveal thickness for any other reason
* Concurrent macular diseases that could confound the results of this study
* Prior vitrectomy in the study eye
* Prior treatment with intravitreal injection including pegaptanib sodium, ranibizumab, bevacizumab or triamcinolone acetonide

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Jumper, M.D., Principal Investigator — West Coast Retina Medical Group, Inc.
Locations (1):
- West Coast Retina Medical Group Inc., San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab: Ranibizumab is being used off-label to test the safety and efficacy of its use in Diabetic Macular Edema post panretinal photocoagulation.
Period: Overall Study
Arm/Group | Ranibizumab
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Pre-PRP Best Corrected Visual Acuity (BCVA) at 3 Months as Expressed as an Early Treatment Diabetic Retinopathy Study (ETDRS) Score (Number of Letters Correctly Read.)
Description: No outcome measures were obtained for this study. Study was terminated by Investigator/Sponsor due to low enrollment. The data was not formally analyzed but reviewed only on a case study basis.
Time Frame: March 2010
Population: 6 subjects were enrolled in the study: 2 in the observation arm and 4 in the treatment arm. There were only 4 visits in the schedule of assessments and 3 of the subjects missed 2 visits or more. Due to the lack of data collected, the mean change in visual acuity could not be accurately analyzed and calculated.
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Mean Change From Pre-PRP Optical Coherence Tomography (OCT) in Central Foveal Thickness and Macular Volume as Assessed by OCT at 1, 2 and 3 Months.
Description: as for outcome 1
Time Frame: March 2010
Population: 6 subjects were enrolled in the study: 2 in the observation arm and 4 in the treatment arm. There were only 4 visits in the schedule of assessments and 3 of the subjects missed 2 visits or more. Due to the lack of data collected, the mean change in central foveal thickness could not be accurately analyzed and calculated.
Groups:
- Ranibizumab: No outcome measures were obtained for this study. Study was terminated by Investigator/Sponsor due to low enrollment. The data was not formally analyzed but reviewed only on a case study basis. Population size was 0.
  Ranibizumab is being used off-label to test the safety and efficacy of its use in Diabetic Macular Edema post panretinal photocoagulation. Ranibizumab 0.5mg at baseline and then again at 30 days and/or 60 days after PRP as deemed appropriate by the Investigator.
  ranibizumab: Ranibizumab 0.5mg at baseline and then again at 30 days and/or 60 days after PRP as deemed appropriate by the Investigator.
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Patients That Maintain Pre-PRP Visual Acuity at the 3 Month Time Point
Description: as for outcome 1
Time Frame: March 2010
Population: 6 subjects were enrolled in the study: 2 in the observation arm and 4 in the treatment arm. There were only 4 visits in the schedule of assessments and 3 of the subjects missed 2 visits or more. Due to the lack of data collected, the percentage of patients that maintain pre-PRP visual acuity could not be accurately analyzed and calculated.
Groups:
- Ranibizumab: No outcome measures were obtained for this study. Study was terminated by Investigator/Sponsor due to low enrollment. The data was not formally analyzed but reviewed only on a case study basis. Population size was 0
  Ranibizumab is being used off-label to test the safety and efficacy of its use in Diabetic Macular Edema post panretinal photocoagulation. Ranibizumab 0.5mg at baseline and then again at 30 days and/or 60 days after PRP as deemed appropriate by the Investigator.
  ranibizumab: Ranibizumab 0.5mg at baseline and then again at 30 days and/or 60 days after PRP as deemed appropriate by the Investigator.
Arm/Group | Ranibizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Study was terminated by Sponsor and Investigator due to low enrollment. Data not analyzed. Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No